CLINICAL TRIAL: NCT01994382
Title: A Phase 1/2a Open-Label, Multi-Dose, Multi-Center Escalation and Exploratory Study of Cerdulatinib (PRT062070) in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) or B-Cell or T-Cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Phase 1/2a Dose Escalation Study in Participants With CLL, SLL, or NHL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-601
Expanded Access: NCT04757259 (No longer available)
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Follicular Lymphoma (FL/Indolent NHL); Aggressive NHL (a NHL); Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL); T-cell Lymphoma (PTCL and CTCL); B-cell Non Hodgkin Lymphoma (NHL)
Keywords: Leukemia; Lymphocytic; Chronic; B Cell
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell; Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell; Leukemia; Bronchiolitis Obliterans Syndrome | interventions — 4-(cyclopropylamino)-2-((4-(4-(ethylsulfonyl)piperazin-1-yl)phenyl)amino)pyrimidine-5-carboxamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1 Cerdulatinib (Experimental): During Phase 1, participants will receive oral cerdulatinib on Day 1 and then starting on Day 4 at doses of 15 mg up to 100 mg QD or oral cerdulatinib at doses of 15 mg up to 45 mg BID in 28-day cycles (except Cohort 1 will have a 21-day cycle starting on Day 1) for up to 10 cycles.
  Interventions: Drug: Cerdulatinib
- Phase 2a Cerdulatinib (Experimental): During Phase 2a, participants in cohorts based on cancer type will receive oral cerdulatinib at starting doses of 35, 30, or 20 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib can be reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID at the discretion of the Investigator based upon clinical judgment and with Sponsor Medical Monitor approval.
  Interventions: Drug: Cerdulatinib
- Phase 2a Cerdulatinib plus Rituximab (Experimental): During Phase 2a, participants in this cohort will receive oral cerdulatinib at their applicable dose and an IV injection of rituximab 375 mg/m^2 on Days 1, 8, 15, and 22 of Cycle 1 and Day 1 of Cycles 4, 6, 8, and 10.
  Interventions: Drug: Cerdulatinib; Biological: Rituximab

INTERVENTIONS:
Drug: Cerdulatinib — Oral capsule
  Other Names: PRT062070; ALXN2075
Biological: Rituximab — IV infusion
  Other Names: Rituxan®; Truxima®; Rixathon®; Ruxience®; MabThera®
  Arms: Phase 2a Cerdulatinib plus Rituximab

SUMMARY:
This study will identify the highest dose, and assess the safety, of cerdulatinib (PRT062070) that may be given in participants with relapsed/refractory chronic lymphocytic leukemia/small lymphocytic lymphoma or non-hodgkin lymphoma.

DETAILED DESCRIPTION:
This is an open-label, Phase 1/2a, multi-dose, multi-center trial of orally administered cerdulatinib assessing safety, tolerability, and pharmacokinetic (PK) parameters conducted in 2 phases:

* Phase 1: Dose-escalation portion, during which participants will be enrolled to receive a single-agent cerdulatinib at their assigned dose level starting at 15 milligrams (mg) once daily (QD), administered in increasing doses until the maximum tolerated dose (MTD)/maximum administered dose (MAD) is identified.
* Phase 2a: Consisting of planned cohorts based on cancer type. The participants will receive single agent cerdulatinib at a starting dose of 35, 30, or 20 mg twice daily (BID) for 28-day cycles except for one of the cohorts, the participants will receive cerdulatinib plus intravenous (IV) rituximab at 375 mg/square meter (m^2) for 28-day cycles.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 Inclusion

• Participant at least 18 years of age with histologically confirmed CLL/SLL or B-cell non-Hodgkin lymphoma (diffuse large B-cell lymphoma [DLBCL], FL, mantle cell lymphoma [MCL], marginal zone lymphoma [MZL], lymphoplasmacytic lymphoma).

Phase 2a Inclusion

* Histological evidence: FL Grade 1-3A, with relapsed or refractory disease; aggressive NHL (aNHL), defined as DLBCL, FL Grade 3B, MCL, and transformed NHL with relapsed disease; CLL/SLL, peripheral T-cell lymphoma (PTCL), or cutaneous T-cell lymphoma (CTCL) (with mycosis fungoides [MF]/Sézary Syndrome [SS]) with relapsed or refractory disease
* Received B-cell receptor (BCR) and/or BCL2 inhibitors and were intolerant or had relapsed/refractory disease afterwards
* Prior treatment for lymphoid malignancy for progressive /refractory disease
* ≥1 prior regimen (minimum 2 cycles) with antibody conjugate/cytotoxic chemotherapy.
* Measurable disease defined as: ≥1 lesion that measures ≥1.5 centimeter (cm) single dimension via computed tomography (CT), CT/positive-emission tomography (PET) with nodal or mass lesions; quantifiable circulating tumor cells; and for CTCL: Modified Severity Weighted Assessment Tool (mSWAT) >0
* Ability to provide diagnostic reports

General Inclusion

* Eastern Cooperative Oncology Group (ECOG) Score of 0 or 1
* Hematologic absolute neutrophil count (ANC) >1000/microliter (uL) and platelet >75,000/uL
* Creatinine levels as specified by Investigator
* Bilirubin <2.0 mg/deciliter [dL] (if Gilberts then <2.5 mg/dL) and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) <2.5*ULN

Exclusion Criteria:

* Richter's syndrome, Burkitt's lymphoma, or Burkitt-like Lymphoma (transformed DLBCL from follicular NHL are eligible)
* Prior transplant with stem cell infusion within 90 days of Day 1 or active graft-versus-host treatment within 8 weeks of Day 1
* Prior therapy with Spleen Tyrosine Kinase (SYK) inhibitors
* Chronic treatment with strong CYP3A4 inhibitor/inducer
* Known lymphomatous involvement of the central nervous system (CNS)
* Persistent, unresolved National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0 ≥Grade 2, previous drug-related toxicity (except alopecia, erectile impotence, hot flashes, libido, neuropathy).
* Prior monoclonal antibody (including alemtuzumab), radioimmunoconjugate, antibody drug conjugate, phototherapy, radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any test agent within 3 weeks of Day 1
* For CTCL: (total skin electron beam therapy [TSEBT]) within 12 weeks, or initiation of topical steroid, nitrogen mustard, or topical retinoid within 2 weeks. Stable topical regimen for ≥4 weeks prior to Day 1 allowed.
* Known carrier or infection for human immunodeficiency virus (HIV)/hepatitis B or C. If hepatitis C virus (HCV) antibody (ab)+, must be polymerase chain reaction (PCR)- to be eligible. If hepatitis B virus (HBV) ab+, must be hepatitis B surface antigen (HBsAg)- or undetectable HBV deoxyribonucleic acid (DNA) to be eligible.
* Active infection requiring systemic treatment,
* Significant gastrointestinal (GI) disease, previous major gastric/bowel surgery, difficulty swallowing, or malabsorption syndrome
* Major surgery within 4 weeks
* Previous malignancies within 2 years unless relapse risk is small (<5%).
* Current use of systemic steroids >20 mg QD prednisone (or equivalent)
* Breastfeeding or pregnant (intention to become) females or participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Portola Study Director, Study Director — Portola Pharmaceuticals
Locations (23):
- United States (23):
  - Huntsville, Alabama
  - Gilbert, Arizona
  - Los Angeles, California
  - Palo Alto, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Sarasota, Florida
  - Lawrenceville, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Hattiesburg, Mississippi
  - Hackensack, New Jersey
  - Morristown, New Jersey
  - New York, New York
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Arlington, Texas
  - Lubbock, Texas
  - Richmond, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Paul A. Hamlin, Manish R. Patel, Don Stevens, Brian T. Hess, Javier Munoz, Tatyana A. Feldman, Sonali M. Smith, Greg P. Coffey, Muhtarjan Osman, Jaymes S Holland, Cristina B Guzman, Stephen D. Smith; Phase 2a Study of the Dual SYK/JAK Inhibitor Cerdulatinib (ALXN2075) As Monotherapy or in Combination with Rituximab in Patients with Relapsed/Refractory Follicular Lymphoma. Blood 2021; 138 (Supplement 1): 2423. doi: https://doi.org/10.1182/blood-2021-148313
- [Derived] Coffey GP, Feng J, Betz A, Pandey A, Birrell M, Leeds JM, Der K, Kadri S, Lu P, Segal J, Wang YL, Michelson G, Curnutte JT, Conley PB. Cerdulatinib Pharmacodynamics and Relationships to Tumor Response Following Oral Dosing in Patients with Relapsed/Refractory B-cell Malignancies. Clin Cancer Res. 2019 Feb 15;25(4):1174-1184. doi: 10.1158/1078-0432.CCR-18-1047. Epub 2018 Oct 17. PMID 30333224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study with 2 phases.
Pre-assignment Details: Phase 1: dose-escalation portion of study, participants received doses of cerdulatinib at assigned regimen. Phase 2a: participants were enrolled into cohorts based on cancer type and received single agent cerdulatinib except for 1 cohort, participants received cerdulatinib+rituximab. Three participants in Phase 1 rolled over to Phase 2; their data are included in respective arms in both phases. Therefore, the data are included twice in the Totals for Participant Flow & Baseline Characteristics.
Groups:
- Phase 1: Cerdulatinib 15 Milligrams (mg) Once Daily (QD): Participants received oral cerdulatinib at 15 mg QD starting on Day 1 in 21-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 30 mg QD: Participants received oral cerdulatinib at 30 mg on Day 1 and then QD starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 45 mg QD: Participants received oral cerdulatinib at 45 mg on Day 1 and then QD starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 15 mg Twice Daily (BID): Participants received oral cerdulatinib at 15 mg on Day 1 and then BID starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 40 mg QD: Participants received oral cerdulatinib at 40 mg on Day 1 and then QD starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 20 mg BID: Participants received oral cerdulatinib at 20 mg on Day 1 and then BID starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 50 mg QD: Participants received oral cerdulatinib at 50 mg on Day 1 and then QD starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 65 mg QD: Participants received oral cerdulatinib at 65 mg on Day 1 and then QD starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 100 mg QD: Participants received oral cerdulatinib at 100 mg on Day 1 and then QD starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 45 mg BID: Participants received oral cerdulatinib at 45 mg on Day 1 and then BID starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 2a: Cerdulatinib (FL Cohort): Participants with follicular lymphoma (FL) received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib (MZL/WM Cohort): Participants with marginal zone lymphoma/Waldenström's macroglobulinemia (MZL/WM) received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort): Participants with FL received oral cerdulatinib at starting doses of 30 or 20 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable. Participants also received intravenous (IV) injections of rituximab 375 milligrams (mg)/square meter (m^2) on Days 1, 8, 15, and 22 of Cycle 1 and Day 1 of Cycles 4, 6, 8, and 10.
- Phase 2a: Cerdulatinib (aNHL Cohort): Participants with aggressive non-Hodgkin lymphoma (aNHL) received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib (CLL/SLL Cohort): Participants with chronic lymphocytic leukemia/small cell lymphocytic lymphoma (CLL/SLL) received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib (PTCL Cohort): Participants with peripheral T-cell lymphoma (PTCL) received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib (CTCL Cohort): Participants with cutaneous T-cell lymphoma (CTCL) received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
Period: Overall Study
Arm/Group | Phase 1: Cerdulatinib 15 Milligrams (mg) Once Daily (QD) | Phase 1: Cerdulatinib 30 mg QD | Phase 1: Cerdulatinib 45 mg QD | Phase 1: Cerdulatinib 15 mg Twice Daily (BID) | Phase 1: Cerdulatinib 40 mg QD | Phase 1: Cerdulatinib 20 mg BID | Phase 1: Cerdulatinib 50 mg QD | Phase 1: Cerdulatinib 65 mg QD | Phase 1: Cerdulatinib 100 mg QD | Phase 1: Cerdulatinib 45 mg BID | Phase 2a: Cerdulatinib (FL Cohort) | Phase 2a: Cerdulatinib (MZL/WM Cohort) | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) | Phase 2a: Cerdulatinib (aNHL Cohort) | Phase 2a: Cerdulatinib (CLL/SLL Cohort) | Phase 2a: Cerdulatinib (PTCL Cohort) | Phase 2a: Cerdulatinib (CTCL Cohort)
Started | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 6 | 3 | 5 | 42 | 12 | 26 | 6 | 28 | 65 | 41
Received at Least 1 Dose of Study Drug (Safety Population) | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 6 | 3 | 5 | 42 | 12 | 26 | 6 | 28 | 65 | 41
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 6 | 3 | 5 | 42 | 12 | 26 | 6 | 28 | 65 | 41
Not completed — Informed consent withdrawn | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 4 | 4 | 3 | 2 | 3 | 3 | 6 | 2 | 2 | 13 | 8 | 7 | 3 | 6 | 44 | 28
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 4 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 2 | 7 | 3 | 17 | 6 | 3
Not completed — Other than specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 2 | 0 | 4 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participants rolled over into expanded access program (NCT04757259) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 0 | 0 | 3 | 2
Not completed — Protocol violation/noncompliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Rolled over to Phase 2a | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Population included participants who received at least 1 dose of study drug.
Groups:
- Phase 1: Cerdulatinib 15 mg QD: Participants received oral cerdulatinib at 15 mg QD starting on Day 1 in 21-day cycles for up to 10 cycles.
- Phase 1: Cerdulatinib 15 mg BID: Participants received oral cerdulatinib at 15 mg on Day 1 and then BID starting on Day 4 in 28-day cycles for up to 10 cycles.
- Phase 2a: Cerdulatinib (FL Cohort): Participants with FL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib (MZL/WM Cohort): Participants with MZL/WM received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort): Participants with FL received oral cerdulatinib at starting doses of 30 or 20 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID. Participants also received IV injections of rituximab 375 mg/m^2 on Days 1, 8, 15, and 22 of Cycle 1 and Day 1 of Cycles 4, 6, 8, and 10.
- Phase 2a: Cerdulatinib (aNHL Cohort): Participants with aNHL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib (CLL/SLL Cohort): Participants with CLL/SLL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib (PTCL Cohort): Participants with PTCL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Phase 2a: Cerdulatinib (CTCL Cohort): Participants with CTCL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Cerdulatinib 15 mg QD | Phase 1: Cerdulatinib 30 mg QD | Phase 1: Cerdulatinib 45 mg QD | Phase 1: Cerdulatinib 15 mg BID | Phase 1: Cerdulatinib 40 mg QD | Phase 1: Cerdulatinib 20 mg BID | Phase 1: Cerdulatinib 50 mg QD | Phase 1: Cerdulatinib 65 mg QD | Phase 1: Cerdulatinib 100 mg QD | Phase 1: Cerdulatinib 45 mg BID | Phase 2a: Cerdulatinib (FL Cohort) | Phase 2a: Cerdulatinib (MZL/WM Cohort) | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) | Phase 2a: Cerdulatinib (aNHL Cohort) | Phase 2a: Cerdulatinib (CLL/SLL Cohort) | Phase 2a: Cerdulatinib (PTCL Cohort) | Phase 2a: Cerdulatinib (CTCL Cohort) | Total
Number analyzed (Participants) | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 6 | 3 | 5 | 42 | 12 | 26 | 6 | 28 | 65 | 41 | 263
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 3 | 0 | 3 | 2 | 0 | 1 | 1 | 1 | 23 | 7 | 13 | 2 | 8 | 33 | 21 | 120
  >=65 years | 2 | 5 | 4 | 3 | 0 | 1 | 4 | 5 | 2 | 4 | 19 | 5 | 13 | 4 | 20 | 32 | 20 | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 2 | 0 | 2 | 1 | 1 | 0 | 2 | 16 | 4 | 9 | 1 | 12 | 24 | 18 | 97
  Male | 3 | 4 | 4 | 1 | 3 | 1 | 3 | 5 | 3 | 3 | 26 | 8 | 17 | 5 | 16 | 41 | 23 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 6 | 1 | 13
  Not Hispanic or Latino | 3 | 6 | 7 | 3 | 3 | 2 | 4 | 6 | 3 | 3 | 37 | 10 | 24 | 5 | 26 | 53 | 37 | 232
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 6 | 3 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 3 | 10 | 11 | 29
  White | 3 | 6 | 7 | 3 | 2 | 3 | 4 | 6 | 3 | 4 | 36 | 11 | 22 | 6 | 23 | 48 | 24 | 211
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 5 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: DLT was defined as any of the following toxicities, possibly or probably related to cerdulatinib, and clinically significant (in the judgement of Investigator): -Febrile neutropenia (absolute neutrophil count <1000/microliter [μL] and temperature ≥38.5°Celcius). -Grade 4 neutropenia for >5 days. -Grade 4 thrombocytopenia with or without bleeding. -Grade 3 thrombocytopenia with bleeding. -Grade 4 anemia, unexplained by underlying disease. -Grade 3 or greater nausea, vomiting, or diarrhea if persistent despite optimal antiemetic or anti-diarrheal therapy. -Grade 3 or greater increase in transaminases lasting >5 days. -Grade 3 or greater fatigue persisting >7 days in absence of any other underlying cause. -Any other Grade 3 or greater non-hematologic toxicity (except fatigue as noted above) considered clinically significant by Investigator. -Toxicity of any grade resulting in dose delay of >7 days. -Toxicity resulting in study drug discontinuation prior to completion of Cycle 1.
Time Frame: Baseline up to Day 28 of Cycle 1 (cycle = 21 days or 28 days)
Population: The Safety Analysis Population included participants who received at least 1 dose of study drug. Only data from participants in Phase 1 cohorts (arms) were applicable and evaluated for this Outcome Measure. Evaluable participants for this Outcome Measure must have received 80% of doses in Cycle 1 or withdrawn from study drug due to drug-related toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Cerdulatinib 15 mg QD | Phase 1: Cerdulatinib 30 mg QD | Phase 1: Cerdulatinib 45 mg QD | Phase 1: Cerdulatinib 15 mg BID | Phase 1: Cerdulatinib 40 mg QD | Phase 1: Cerdulatinib 20 mg BID | Phase 1: Cerdulatinib 50 mg QD | Phase 1: Cerdulatinib 65 mg QD | Phase 1: Cerdulatinib 100 mg QD | Phase 1: Cerdulatinib 45 mg BID
Number analyzed (Participants) | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 6 | 3 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

2. Primary Outcome: Phase 2a: Number of Participants Achieving Overall Response Rate (Partial Response [PR] Plus Complete Response [CR]) as Assessed by the Investigator
Description: CR included: -Via a positron emission tomography (PET)/computed tomography (CT) scan, score of 1 (no uptake above background), 2 (uptake of <mediastinum), or 3 (uptake of >mediastinum but <liver) for lymph nodes and extralymphatic sites; no new lesions; and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. -Via CT scan, target nodes/nodal masses regressed to <1.5 centimeters (cm) in longest transverse diameter of a lesion (LDi); no extralymphatic sites of disease; organ enlargement has regressed to normal; and bone marrow was normal by morphology and if indeterminate, immunohistochemistry was negative.
  PR included: -Via a PET/CT scan, score of 4 (uptake of moderately >liver) or 5 (uptake markedly higher than liver and/or new lesions) with reduced uptake compared with baseline and residual masses of any size. -Via CT scan, >50% decrease in the sum of the product of perpendicular diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites.
Time Frame: Baseline up to End of Treatment (up to last day of Cycle 10 [cycle = 28 days])
Population: The Efficacy Analysis Population included all participants who took at least 1 dose of study drug and had at least 1 post-baseline Investigator response assessment. Only the cohorts (arms) with participants with FL or with PTCL were applicable and evaluated for this Outcome Measure. Here, 'Number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2a: Cerdulatinib (FL Cohort) With ≤3 Prior Regimen: Participants with FL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable. Participants in this cohort received prior treatment regimen of ≤3 times before study start.
- Phase 2a: Cerdulatinib (FL Cohort) With ≥4 Prior Regimen: Participants with FL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable. Participants in this cohort received prior treatment regimen of ≥4 times before study start.
- Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≤3 Prior Regimen: Participants with FL received oral cerdulatinib at starting doses of 30 or 20 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable. Participants also received IV injections of rituximab 375 mg/m^2 on Days 1, 8, 15, and 22 of Cycle 1 and Day 1 of Cycles 4, 6, 8, and 10. Participants in this cohort received prior treatment regimen of ≤3 times before study start.
- Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≥4 Prior Regimen: Participants with FL received oral cerdulatinib at starting doses of 30 or 20 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable. Participants also received IV injections of rituximab 375 mg/m^2 on Days 1, 8, 15, and 22 of Cycle 1 and Day 1 of Cycles 4, 6, 8, and 10. Participants in this cohort received prior treatment regimen of ≥4 times before study start.
- Phase 2a: Cerdulatinib (PTCL Cohort) With AITL/TFH: Participants with PTCL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable. This cohort included participants with cancer type of PTCL angioimmunoblastic T-cell lymphoma (AITCL/AITL) and PTCL with T-follicular helper phenotype (TFH).
- Phase 2a: Cerdulatinib (PTCL Cohort) With NOS: Participants with PTCL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable. This cohort included participants with cancer type of PTCL not otherwise specified (NOS).
- Phase 2a: Cerdulatinib (PTCL Cohort) With Other: Participants with PTCL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable. This cohort included participants with cancer type of other PTCL pathology subgroups not included in AITL/TFH or NOS subgroups.
Arm/Group | Phase 2a: Cerdulatinib (FL Cohort) With ≤3 Prior Regimen | Phase 2a: Cerdulatinib (FL Cohort) With ≥4 Prior Regimen | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≤3 Prior Regimen | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≥4 Prior Regimen | Phase 2a: Cerdulatinib (PTCL Cohort) With AITL/TFH | Phase 2a: Cerdulatinib (PTCL Cohort) With NOS | Phase 2a: Cerdulatinib (PTCL Cohort) With Other
Number analyzed (Participants) | 24 | 10 | 16 | 10 | 27 | 9 | 22
Participants | 12 | 6 | 15 | 5 | 14 | 0 | 7

3. Secondary Outcome: Phase 1: Number of Participants Achieving Overall Response Rate (Partial Response [PR] Plus Complete Response [CR]) as Assessed by the Investigator
Description: CR included: -Via a PET/CT scan, score of 1 (no uptake above background), 2 (uptake of <mediastinum), or 3 (uptake of >mediastinum but <liver) for lymph nodes and extralymphatic sites; no new lesions; and no evidence of FDG-avid disease in bone marrow. -Via CT scan, target nodes/nodal masses regressed to <1.5 cm in LDi; no extralymphatic sites of disease; organ enlargement has regressed to normal; and bone marrow was normal by morphology and if indeterminate, immunohistochemistry was negative.
  PR included: -Via a PET/CT scan, a score of 4 (uptake of moderately >liver) or 5 (uptake markedly higher than liver and/or new lesions) with reduced uptake compared with baseline and residual masses of any size. -Via CT scan, >50% decrease in the sum of the product of perpendicular diameters for multiple lesion of up to 6 target measurable nodes and extranodal sites.
Time Frame: Baseline up to End of Treatment (up to last day of Cycle 10 [cycle = 21 days or 28 days])
Population: The Safety Analysis Population included participants who received at least 1 dose of study drug. Only data from participants in Phase 1 cohorts (arms) were applicable and evaluated for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Cerdulatinib 15 mg QD | Phase 1: Cerdulatinib 30 mg QD | Phase 1: Cerdulatinib 45 mg QD | Phase 1: Cerdulatinib 15 mg BID | Phase 1: Cerdulatinib 40 mg QD | Phase 1: Cerdulatinib 20 mg BID | Phase 1: Cerdulatinib 50 mg QD | Phase 1: Cerdulatinib 65 mg QD | Phase 1: Cerdulatinib 100 mg QD | Phase 1: Cerdulatinib 45 mg BID
Number analyzed (Participants) | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 6 | 3 | 5
Participants | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2

4. Secondary Outcome: Phase 1: Number of Participants Achieving Clinical Benefit
Description: Clinical benefit was defined as achieving stable disease (SD) or better, as assessed by the Investigator. SD included: -Via a PET/CT scan, a score of 4 (uptake of moderately >liver) or 5 (uptake markedly higher than liver and/or new lesions) with no significant change in FDG uptake from baseline at interim or end of treatment; no new lesions; and no change from baseline in bone marrow. -Via CT scan, <50% decrease from baseline in sum of products of the greatest perpendicular diameters (SPD) of up to 6 dominant, measurable nodes and extranodal sites; no increase consistent with progression in nonmeasured lesions or organ enlargement; and no new lesions.
Time Frame: Baseline up to End of Treatment (up to last day of Cycle 10 [cycle = 21 days or 28 days])
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Cerdulatinib 15 mg QD | Phase 1: Cerdulatinib 30 mg QD | Phase 1: Cerdulatinib 45 mg QD | Phase 1: Cerdulatinib 15 mg BID | Phase 1: Cerdulatinib 40 mg QD | Phase 1: Cerdulatinib 20 mg BID | Phase 1: Cerdulatinib 50 mg QD | Phase 1: Cerdulatinib 65 mg QD | Phase 1: Cerdulatinib 100 mg QD | Phase 1: Cerdulatinib 45 mg BID
Number analyzed (Participants) | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 6 | 3 | 5
Participants | 2 | 4 | 4 | 1 | 1 | 0 | 2 | 2 | 1 | 1

5. Secondary Outcome: Phase 1 and Phase 2: Number of Participants With an Adverse Event (AE) or a Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence, which may or may not have a causal relationship to the study drug, including: unfavorable and unintended sign, symptom, or disease temporally associated with the use of the study drug; any newly occurring event or exacerbation of previous condition (for example, increase in severity or frequency) since the administration of study drug; recurrence of an intermittent medical condition not present at baseline; any deterioration in a laboratory value or other clinical test that is associated with symptoms or leads to a change in study treatment or concomitant treatment or discontinuation from study drug; and AEs related to a study intervention. An SAE is an AE that is fatal, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or a congenital anomaly/birth defect.
Time Frame: Baseline up to End of Study (up to 30 days after last dose in Cycle 10 [cycle = up to 28 days])
Population: The Safety Analysis Population included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2a: Cerdulatinib (FL Cohort): Participants with FL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable, at the discretion of the Investigator based upon clinical judgment and with Sponsor Medical Monitor approval.
- Phase 2a: Cerdulatinib (MZL/WM Cohort): Participants with MZL/WM received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable, at the discretion of the Investigator based upon clinical judgment and with Sponsor Medical Monitor approval.
- Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort): Participants with FL received oral cerdulatinib at starting doses of 30 or 20 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable, at the discretion of the Investigator based upon clinical judgment and with Sponsor Medical Monitor approval. Participants also received IV injections of rituximab 375 mg/m^2 on Days 1, 8, 15, and 22 of Cycle 1 and Day 1 of Cycles 4, 6, 8, and 10.
- Phase 2a: Cerdulatinib (aNHL Cohort): Participants with aNHL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable, at the discretion of the Investigator based upon clinical judgment and with Sponsor Medical Monitor approval.
- Phase 2a: Cerdulatinib (CLL/SLL Cohort): Participants with CLL/SLL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable, at the discretion of the Investigator based upon clinical judgment and with Sponsor Medical Monitor approval.
- Phase 2a: Cerdulatinib (PTCL Cohort): Participants with PTCL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable, at the discretion of the Investigator based upon clinical judgment and with Sponsor Medical Monitor approval.
- Phase 2a: Cerdulatinib (CTCL Cohort): Participants with CTCL received oral cerdulatinib at starting doses of 35 or 30 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable, at the discretion of the Investigator based upon clinical judgment and with Sponsor Medical Monitor approval.
Arm/Group | Phase 1: Cerdulatinib 15 mg QD | Phase 1: Cerdulatinib 30 mg QD | Phase 1: Cerdulatinib 45 mg QD | Phase 1: Cerdulatinib 15 mg BID | Phase 1: Cerdulatinib 40 mg QD | Phase 1: Cerdulatinib 20 mg BID | Phase 1: Cerdulatinib 50 mg QD | Phase 1: Cerdulatinib 65 mg QD | Phase 1: Cerdulatinib 100 mg QD | Phase 1: Cerdulatinib 45 mg BID | Phase 2a: Cerdulatinib (FL Cohort) | Phase 2a: Cerdulatinib (MZL/WM Cohort) | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) | Phase 2a: Cerdulatinib (aNHL Cohort) | Phase 2a: Cerdulatinib (CLL/SLL Cohort) | Phase 2a: Cerdulatinib (PTCL Cohort) | Phase 2a: Cerdulatinib (CTCL Cohort)
Number analyzed (Participants) | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 6 | 3 | 5 | 42 | 12 | 26 | 6 | 28 | 65 | 41
Participants
  AE | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 6 | 3 | 5 | 42 | 12 | 26 | 6 | 28 | 65 | 41
  SAE | 0 | 2 | 4 | 0 | 1 | 0 | 2 | 2 | 2 | 3 | 22 | 2 | 7 | 3 | 17 | 42 | 21

6. Secondary Outcome: Phase 1: Area Under the Plasma Concentration-Time Curve From 0 to 12 Hours (AUC0-12) of Cerdulatinib
Time Frame: Cycle (C)1 Day (D)1: predose (0), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, and 72 hours postdose (except 15mg QD); C1D1: 0, 0.5, 1, 2, 3, 4, 6, 8, and 12 hours postdose (15mg QD); C2D1: 0, 0.5, 1, 2, 3, 4, 6, 8, and 12 hours postdose (all doses)
Population: The Pharmacokinetic Analysis Population consisted of all participants who received the requisite treatments and have data at the required timepoints. Only data from participants in Phase 1 cohorts (arms) were applicable and evaluated for this Outcome Measure. Here, 'Number of participants analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: hours*nanograms/milliliter (h*ng/mL)
Arm/Group | Phase 1: Cerdulatinib 15 mg QD | Phase 1: Cerdulatinib 30 mg QD | Phase 1: Cerdulatinib 45 mg QD | Phase 1: Cerdulatinib 15 mg BID | Phase 1: Cerdulatinib 40 mg QD | Phase 1: Cerdulatinib 20 mg BID | Phase 1: Cerdulatinib 50 mg QD | Phase 1: Cerdulatinib 65 mg QD | Phase 1: Cerdulatinib 100 mg QD | Phase 1: Cerdulatinib 45 mg BID
Number analyzed (Participants) | 3 | 6 | 7 | 3 | 3 | 3 | 4 | 5 | 3 | 5
hours*nanograms/milliliter (h*ng/mL)
  Day 1 of Cycle 1 | 709.6 (37.823) | 1040 (347.34) | 1826 (713.67) | 601.4 (118.04) | 2064 (666.52) | 674.5 (113.34) | 2465 (305.70) | 2719 (1208.2) | 2758 (969.37) | 1335 (530.56)
  Day 1 of Cycle 2: number analyzed (Participants) | 3 | 6 | 6 | 3 | 2 | 2 | 3 | 3 | 0 | 0
  Day 1 of Cycle 2 | 1321 (140.21) | 1900 (918.79) | 6804 (3065.6) | 2129 (533.14) | 6313 (166.81) | 2779 (458.94) | 5871 (3685.1) | 6215 (249.64) |  |

7. Secondary Outcome: Phase 2a: Median Time to Progression-Free Survival (PFS)
Description: PFS=(first documentation of disease progression [DP] or death [whichever occurred first]-study drug first dose date+1)/30.4375 in months. PFS right censored for 1 of these conditions: 1) no baseline disease assessments; 2) starting new anticancer therapy before documented DP/death; 3) DP/death immediately after >6 months since last disease assessment (or >12 months if after last cycle); & alive without documented DP. 95% confidence interval estimated using Brookmeyer method. DP included: -Via a PET/CT scan, score of 4 (uptake of moderately >liver) or 5 (uptake markedly higher than liver and/or new lesions) with uptake increase in intensity, new FDG-avid foci, & no nonmeasured lesions. -Via CT, abnormal individual node/lesion with significant LDi or shortest axis perpendicular to LDi increase; prior splenomegaly, >50% splenic length increase; if no prior splenomegaly, ≥2 cm splenic length increase; new or recurrent splenomegaly; new/clear progression of preexisting nonmeasured lesions.
Time Frame: Baseline up to End of Treatment (up to last day of Cycle 10 [cycle = 28 days])
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2a: Cerdulatinib (FL Cohort) With ≤3 Prior Regimen | Phase 2a: Cerdulatinib (FL Cohort) With ≥4 Prior Regimen | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≤3 Prior Regimen | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≥4 Prior Regimen | Phase 2a: Cerdulatinib (PTCL Cohort) With AITL/TFH | Phase 2a: Cerdulatinib (PTCL Cohort) With NOS | Phase 2a: Cerdulatinib (PTCL Cohort) With Other
Number analyzed (Participants) | 24 | 10 | 16 | 10 | 27 | 9 | 22
months | 12.68 [4.53 to NA] — NA=not applicable. Due to several participants who were censored (see conditions detailed above) the upper limit could not be estimated. | 3.61 [1.28 to NA] — Due to several participants who were censored (see conditions detailed above) the upper limit could not be estimated. | 18.33 [10.74 to NA] — Due to several participants who were censored (see conditions detailed above) the upper limit could not be estimated. | NA [3.58 to NA] — Due to several participants who were censored (see conditions detailed above) the median and the upper limit could not be estimated. | 4.57 [1.71 to 9.99] | 1.18 [0.26 to 3.58] | 3.45 [2.07 to 5.62]

8. Secondary Outcome: Phase 2a: Number of Participants Achieving Clinical Benefit
Description: Clinical benefit was defined as achieving SD or better, as assessed by the Investigator. SD included: -Via a PET/CT scan, a score of 4 (uptake of moderately >liver) or 5 (uptake markedly higher than liver and/or new lesions) with no significant change in FDG uptake from baseline at interim or end of treatment; no new lesions; and no change from baseline in bone marrow. -Via CT scan, <50% decrease from baseline in sum of products of the greatest perpendicular diameters (SPD) of up to 6 dominant, measurable nodes and extranodal sites; no increase consistent with progression in nonmeasured lesions or organ enlargement; and no new lesions.
Time Frame: Baseline up to End of Treatment (up to last day of Cycle 10 [cycle = 28 days])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a: Cerdulatinib (FL Cohort) With ≤3 Prior Regimen | Phase 2a: Cerdulatinib (FL Cohort) With ≥4 Prior Regimen | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≤3 Prior Regimen | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≥4 Prior Regimen | Phase 2a: Cerdulatinib (PTCL Cohort) With AITL/TFH | Phase 2a: Cerdulatinib (PTCL Cohort) With NOS | Phase 2a: Cerdulatinib (PTCL Cohort) With Other
Number analyzed (Participants) | 24 | 10 | 16 | 10 | 27 | 9 | 22
Participants | 19 | 8 | 16 | 10 | 17 | 2 | 16

9. Secondary Outcome: Phase 2a: Number of Participants Achieving Dominant Mass Response (DMR)
Description: DMR was defined as achieving a ≥50% decrease from baseline in the SPD of the target nodal and extranodal lesions. SPD at a visit was considered missing if any target lesion was not evaluated.
Time Frame: Baseline up to End of Treatment (up to last day of Cycle 10 [cycle = 28 days])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a: Cerdulatinib (FL Cohort) With ≤3 Prior Regimen | Phase 2a: Cerdulatinib (FL Cohort) With ≥4 Prior Regimen | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≤3 Prior Regimen | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) With ≥4 Prior Regimen | Phase 2a: Cerdulatinib (PTCL Cohort) With AITL/TFH | Phase 2a: Cerdulatinib (PTCL Cohort) With NOS | Phase 2a: Cerdulatinib (PTCL Cohort) With Other
Number analyzed (Participants) | 24 | 10 | 16 | 10 | 27 | 9 | 22
Participants | 14 | 5 | 14 | 7 | 15 | 1 | 5

ADVERSE EVENTS:
Time Frame: Baseline up to End of Study (up to 30 days after last dose in Cycle 10 [cycle = up to 28 days])
Description: The Safety Analysis Population included participants who received at least 1 dose of study drug.
Groups:
- Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort): Participants with FL received oral cerdulatinib at starting doses of 30 or 20 mg BID on Day 1 in 28-day cycles for up to 10 cycles. Doses of cerdulatinib could have been reduced to a minimum dose of 15 mg BID or increased to a maximum dose of 30 mg BID, when applicable. Participants also received IV injections of rituximab 375 mg/m^2 on Days 1, 8, 15, and 22 of Cycle 1 and Day 1 of Cycles 4, 6, 8, and 10.
Arm/Group | Phase 1: Cerdulatinib 15 mg QD | Phase 1: Cerdulatinib 30 mg QD | Phase 1: Cerdulatinib 45 mg QD | Phase 1: Cerdulatinib 15 mg BID | Phase 1: Cerdulatinib 40 mg QD | Phase 1: Cerdulatinib 20 mg BID | Phase 1: Cerdulatinib 50 mg QD | Phase 1: Cerdulatinib 65 mg QD | Phase 1: Cerdulatinib 100 mg QD | Phase 1: Cerdulatinib 45 mg BID | Phase 2a: Cerdulatinib (FL Cohort) | Phase 2a: Cerdulatinib (MZL/WM Cohort) | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) | Phase 2a: Cerdulatinib (aNHL Cohort) | Phase 2a: Cerdulatinib (CLL/SLL Cohort) | Phase 2a: Cerdulatinib (PTCL Cohort) | Phase 2a: Cerdulatinib (CTCL Cohort)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/7 | 0/3 | 1/3 | 0/3 | 0/4 | 0/6 | 1/3 | 1/5 | 0/42 | 0/12 | 0/26 | 0/6 | 0/28 | 1/65 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/6 | 4/7 | 0/3 | 1/3 | 0/3 | 2/4 | 2/6 | 2/3 | 3/5 | 22/42 | 2/12 | 7/26 | 3/6 | 17/28 | 42/65 | 21/41
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 7/7 | 3/3 | 3/3 | 3/3 | 4/4 | 6/6 | 3/3 | 5/5 | 42/42 | 12/12 | 26/26 | 6/6 | 28/28 | 65/65 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Cerdulatinib 15 mg QD (N=3) | Phase 1: Cerdulatinib 30 mg QD (N=6) | Phase 1: Cerdulatinib 45 mg QD (N=7) | Phase 1: Cerdulatinib 15 mg BID (N=3) | Phase 1: Cerdulatinib 40 mg QD (N=3) | Phase 1: Cerdulatinib 20 mg BID (N=3) | Phase 1: Cerdulatinib 50 mg QD (N=4) | Phase 1: Cerdulatinib 65 mg QD (N=6) | Phase 1: Cerdulatinib 100 mg QD (N=3) | Phase 1: Cerdulatinib 45 mg BID (N=5) | Phase 2a: Cerdulatinib (FL Cohort) (N=42) | Phase 2a: Cerdulatinib (MZL/WM Cohort) (N=12) | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) (N=26) | Phase 2a: Cerdulatinib (aNHL Cohort) (N=6) | Phase 2a: Cerdulatinib (CLL/SLL Cohort) (N=28) | Phase 2a: Cerdulatinib (PTCL Cohort) (N=65) | Phase 2a: Cerdulatinib (CTCL Cohort) (N=41)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 3 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 5 | 0 | 4 | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 5 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Hodgkin lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Nocardiosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corynebacterium sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytomegalovirus gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scedosporium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
West Nile viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fistula of small intestine (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uvulitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 2
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acute motor axonal neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Cerdulatinib 15 mg QD (N=3) | Phase 1: Cerdulatinib 30 mg QD (N=6) | Phase 1: Cerdulatinib 45 mg QD (N=7) | Phase 1: Cerdulatinib 15 mg BID (N=3) | Phase 1: Cerdulatinib 40 mg QD (N=3) | Phase 1: Cerdulatinib 20 mg BID (N=3) | Phase 1: Cerdulatinib 50 mg QD (N=4) | Phase 1: Cerdulatinib 65 mg QD (N=6) | Phase 1: Cerdulatinib 100 mg QD (N=3) | Phase 1: Cerdulatinib 45 mg BID (N=5) | Phase 2a: Cerdulatinib (FL Cohort) (N=42) | Phase 2a: Cerdulatinib (MZL/WM Cohort) (N=12) | Phase 2a: Cerdulatinib Plus Rituximab (FL Cohort) (N=26) | Phase 2a: Cerdulatinib (aNHL Cohort) (N=6) | Phase 2a: Cerdulatinib (CLL/SLL Cohort) (N=28) | Phase 2a: Cerdulatinib (PTCL Cohort) (N=65) | Phase 2a: Cerdulatinib (CTCL Cohort) (N=41)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 2 | 2 | 0 | 2 | 4 | 3 | 5 | 23 | 5 | 21 | 2 | 20 | 27 | 20
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 2 | 2 | 0 | 2 | 0 | 2 | 23 | 6 | 13 | 3 | 14 | 21 | 17
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 3 | 2 | 1 | 13 | 2 | 7 | 1 | 6 | 16 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 10 | 2 | 8 | 2 | 2 | 4 | 6
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 9 | 2 | 6 | 3 | 6 | 6 | 5
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 1 | 1 | 4 | 2
Fatigue (General disorders) | 0 | 2 | 6 | 0 | 1 | 1 | 2 | 5 | 1 | 3 | 21 | 7 | 15 | 2 | 16 | 18 | 14
Pyrexia (General disorders) | 0 | 2 | 4 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 12 | 1 | 5 | 1 | 6 | 8 | 4
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 7 | 1 | 5 | 2 | 11 | 8 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 2 | 4 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 7 | 2 | 4 | 0 | 9 | 6 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 9 | 1 | 4 | 1 | 5 | 8 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 0 | 2 | 1 | 4 | 7 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 5 | 1 | 9 | 4 | 1
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 0 | 2 | 1 | 3 | 10 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 4 | 4 | 6 | 2 | 9 | 21 | 12
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 8 | 0 | 4 | 13 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 2 | 3
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 11 | 2 | 4 | 1 | 7 | 12 | 3
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 1 | 2 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 11 | 0 | 2 | 0 | 4 | 8 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 7 | 0 | 3 | 0 | 2 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 3 | 0 | 4 | 7 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 4 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 5 | 0 | 1 | 8 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 4 | 1 | 3 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 1 | 3
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 2 | 0 | 3 | 4 | 4
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 0 | 4 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 1 | 0 | 2 | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 4 | 7 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 4 | 5 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 1 | 1 | 2
Lipase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 3 | 10 | 0 | 8 | 19 | 24
Amylase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 2 | 7 | 0 | 6 | 28 | 21
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 1 | 1 | 5 | 7
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 10 | 5
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 1 | 4 | 4
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 7
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 4 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 1 | 2 | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 3 | 0 | 4 | 3 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 3 | 3 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 4 | 1 | 7 | 13 | 8
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 5 | 1 | 8 | 6 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 4 | 2 | 4
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 4 | 1 | 4 | 3 | 5
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 4 | 2 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 1 | 8 | 1 | 4 | 3 | 3

LIMITATIONS AND CAVEATS:
Key limitations of the study included that it was originally a single-arm, short-term study; disease progression was included as an AE; inadequate follow-up for death or progression; a lack of use of antimicrobial prophylaxis; and no uniform gastrointestinal toxicity management algorithm. These limitations impacted dose reduction and discontinuations due to treatment emergent AEs. In addition, monitoring issues due to the COVID-19 pandemic also factored into data collection and verification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT01994382/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT01994382/SAP_001.pdf